CLINICAL TRIAL: NCT00905918
Title: A Randomized Study to Investigate the Presence of Tocopherol Metabolites in the Colon
Brief Title: Vitamin E Supplements in Treating Patients Undergoing Surgery for Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120901; CDR0000642446 (Other: NIH); 0220090065 (Other: IRB); P30CA072720 (NIH)
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (No Intervention): Patients receive no intervention before undergoing planned surgery.
- Arm II (Experimental): Patients receive oral high γ-tocopherol vitamin E mixture supplementation once daily for 1 week before undergoing planned surgery.
  Interventions: Dietary Supplement: vitamin E; Other: laboratory biomarker analysis
- Arm III (Experimental): Patients receive oral high γ-tocopherol vitamin E mixture supplementation once daily for 2 weeks before undergoing planned surgery.
  Interventions: Dietary Supplement: vitamin E; Other: laboratory biomarker analysis

INTERVENTIONS:
Dietary Supplement: vitamin E — Given orally
  Arms: Arm II; Arm III
Other: laboratory biomarker analysis — All patients undergo biomarker analyses
  Arms: Arm II; Arm III

SUMMARY:
RATIONALE: Vitamin E may help prevent the development of cancer. Studying samples of tissue from patients with colorectal cancer who receive Vitamin E before undergoing surgery in the laboratory may help doctors learn more about how Vitamin E changes biomarkers related to colorectal cancer.

PURPOSE: This randomized early phase I trial is studying giving vitamin E supplements to see how it affects biomarkers in patients undergoing surgery for colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of high γ-tocopherol vitamin E mixture supplementation on plasma levels of α-, γ-, and δ-tocopherols, and prostaglandin E_2 in patients planning to undergo surgery for colorectal cancer by comparing the blood samples collected before and after the supplementation in each of the groups and analyzing levels of tocopherols and their metabolites in urine samples.
* Test the hypothesis that the supplementation reduces oxidative and nitrosative stress by measuring plasma levels of F_2-isoprostane, C-reactive protein, and 3-nitrotyrosine as well as urinary levels of 8-hydroxy-2-deoxyguanosine (8-OHdG).
* Determine the levels of α-, γ-, and δ-tocopherols in colon tissues and analyze immunohistochemically for cell proliferation, apoptosis, β-catenin localization, RXR expression, cyclooxygenase-2, 8-OHdG, and 3-nitrotyrosine levels in colon cancer tissue slides.

OUTLINE: This is a multicenter study. The first 5 patients receive no supplements (to establish laboratory standards), all other patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive no intervention before undergoing planned surgery.
* Arm II: Patients receive oral high γ-tocopherol vitamin E mixture supplementation once daily for 1 week before undergoing planned surgery.
* Arm III: Patients receive oral high γ-tocopherol vitamin E mixture supplementation once daily for 2 weeks before undergoing planned surgery.

Blood and urine samples are collected at baseline and on the day of surgery for tocopherol and biomarker analysis. A sample of colon tissue is removed during standard surgical resection for chemical analysis. Plasma, tumor tissue, and nontumorous tissues are analyzed for levels of F_2-isoprostane, 8-OHdG, 3-nitrotyrosine, and prostaglandin E_2 via enzyme immunoassays and for levels of α-, γ-, and δ-tocopherols via HPLC.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Suspected or confirmed colorectal cancer meeting the following criteria:

  * Scheduled for surgery as the initial treatment
  * Referred to the Cancer Institute of New Jersey or the Robert Wood Johnson University Hospital
* No requirement for urgent surgery (i.e., surgery that cannot wait for 2 weeks)

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Patients deemed in adequate health to undergo colon resection by their surgeon
* No uncontrolled diabetes, uncontrolled BP, chronic congestive heart failure, or history of renal insufficiency
* No personal or family history of bleeding disorders
* No known history of problems absorbing fats (e.g., Crohn disease, cystic fibrosis)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy for the treatment of this cancer
* More than 2 weeks since prior NSAIDs or corticosteroids
* No concurrent colestipol or orlistat
* No concurrent warfarin or dicumarol
* No concurrent supplementation of vitamin E

  * A multivitamin containing ≤ 60 IU vitamin E allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Plasma and urine levels of α-, γ-, and δ-tocopherols, and prostaglandin E2 | 4 years
Plasma levels of F2-isoprostane, C-reactive protein, and 3-nitrotyrosine and urinary levels of 8-hydroxy-2-deoxyguanosine (8-OHdG) | 4 years
Presence in colon tissue of α-, γ-, and δ-tocopherols, cell proliferation and apoptosis indicators, β-catenin localization, RXR expression, and cyclooxygenase-2, 8-OHdG, and 3-nitrotyrosine levels | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Goodin, PharmD, FCCP, BCOP, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States